CLINICAL TRIAL: NCT06881420
Title: A Prospective Multicenter Registry Study on BASIS Technique for Endovascular Therapy of Acute Large Vessel Occlusion Strokes Due to Intracranial Atherosclerotic Disease (BASIS-DUO)
Brief Title: A Prospective Multicenter Registry Study on BASIS Technique for Endovascular Therapy of Acute Large Vessel Occlusion Strokes Due to Intracranial Atherosclerotic Disease
Status: Recruiting | Type: Observational
Sponsor: Fujian Medical University Union Hospital (Other)
Collaborators: Zhangzhou Municipal Hospital of Fujian Province (Other); First Affiliated Hospital of Jinan University (Other)
Responsible Party: Sponsor
Other Study IDs: FujianUnionHospital
Record Dates: First submitted 2025-01-19; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-01

CONDITIONS: Acute Ischemic Stroke; ICAS - Intracranial Atherosclerosis
Keywords: Acute Ischemic Stroke; ICAS - Intracranial Atherosclerosis; Endovascular thrombectomy; BASIS
MeSH Terms: conditions — Ischemic Stroke; Intracranial Arteriosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- using BASIS technique
  Interventions: Procedure: BASIS technique

INTERVENTIONS:
Procedure: BASIS technique — Balloon AngioplaSty with the dIstal protection of Stent retriever

SUMMARY:
This study will explore the safety and efficacy of BASIS technology in ICAS-LVO lesions through a multicenter, prospective, registry, observational single-arm study.By registering intraoperative recanalization using this technique time, recanalization grade, operative thrombectomy times, intraoperative complications perforating branch occlusion, vascular dissection, vascular rupture, Ectopic thrombus, probability of symptomatic intracranial hemorrhage, mRS Score and mortality rate were followed up for 3 months The unique advantages of the application of the assessment BASIS in this type of lesion provide new insights into complex lesions such as ICAS-LVO The thought and operation method can shorten the operation time, improve the good prognosis, reduce the economic burden and reduce the operation Complications make a positive contribution to ensure that patients receive safe, effective and precise treatment.

DETAILED DESCRIPTION:
This project intends to set up a prospective multi-center single-arm study with no control group and no upper limit of cases.

Using BASIS (Balloon AngioplaSty with the dIstal protection of Stent retriever) technique .

- Balloon angioplasty under the protection of the remote thrombectomy stent for intravascular treatment, such as the BASIS technique for thrombectomy loss Failure, the surgeon can take different techniques for remedial treatment.

1. Construct the three-axis system and establish the path. The microcatheter passes 15mm through the distal end of the thrombus Above, after the thrombectomy stent covering the narrow segment was released, angiography was performed to observe the stenosis and distal thrombus.
2. Use the anchoring effect of the thrombectomy bracket to pull the microcatheter out of the body.
3. Send the guide wire along the thrombectomy stent to the balloon expansion catheter, and place the balloon in the narrow section. At this time, follow the blood The position of the plug relative to the stenosis determines whether to semi-retrieve the Syphonet® plug holder, fill the balloon for expansion, Balloon pressure relief.
4. Use the distal end of the thrombectomy stent to anchor and the support of the balloon dilating catheter to advance the thrombectomy catheter.

   Until the end of the thrombus suction catheter reaches the narrow site.
5. Remove the balloon to enlarge the suction cavity and remove the thrombus using SWIM technique.
6. The residual thrombus was cleaned up and the thrombectomy stent was released again. The thrombectomy stent was recovered after angiographic observation: assembled in vitro With the microcatheter, the thrombectomy stent was released again via the microcatheter. Angiography was performed to observe the treatment of thrombus and stenosis Avoid thrombus escape due to direct hand angiography, if there is still thrombus, continue mechanical thrombus removal until the thrombus is cleared After the microcatheter was recovered and the thrombectomy scaffold was withdrawn, the micro

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old;
* Ischemic stroke;
* Within 72 hours from the onset of symptoms to the time of visit, including post-awakening stroke or blindness For stroke patients, the time when symptoms start is defined as "the last normal time";
* Neuroimaging examination indicated occlusion of anterior or posterior intracranial large vessels, TOAST type was large atherosclerosis type.
* BASIS technique was used for intravascular therapy.

Exclusion Criteria:

* Neuroimaging findings on admission, acute occlusion of multiple vessels and tandem lesions;
* History of atrial fibrillation or heart valve surgery;
* There are clinical contraindications to the use of antiplatelet drugs (hemophilia or thrombocytopenia).Rare disease, known history of coagulation disorders, platelet abnormalities; There is active internal bleeding, intracranial Bleeding history, arteriovenous malformation, aneurysm, etc.);
* Other types of stroke, including hemorrhagic stroke.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICAS-LAO stroke
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
mRS scores at 90 days | 90 days
  functional recovery, assessed by change in modified Rankin Scale (mRS) scores (ranging from 0 [no symptoms] to 6 [death]) at 90 days after onset
FPE:first pass effect | From enrollment to the end of the surgery about 3 hours
  Vascular revascularization rate by basis technique at the first attempt

SECONDARY OUTCOMES:
Residual stenosis rate of target vessel | From enrollment to the end of the surgery about 3 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided